CLINICAL TRIAL: NCT06702904
Title: Evaluation of Neuroprosthesis with Sensory Feedback for Modulation of Phantom Limb Pain and Enhancing Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Skolkovo Institute of Science and Technology (Other)
Collaborators: Motorica LLC (Unknown); The Federal Center of Brain Research and Neurotechnologies (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Skoltech-CNBR5
Record Dates: First submitted 2024-11-13; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Phantom Limb Pain
Keywords: Neuromodulation; Phantom limb pain; Neuropathic pain; Neurostimulation; Chronic pain; Peripheral nerve stimulation; PNS; Spinal cord stimulation; SCS; Dorsal root ganglion stimulation; DRG; Cortical stimulation; Amputation; Neurotechnology; Neuroprosthetics; BCI
MeSH Terms: conditions — Phantom Limb; Neuralgia; Chronic Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Peripheral nerve stimulation for upper-limb prosthesis (Experimental)
  Interventions: Procedure: Peripheral Nerve Stimulation
- Peripheral nerve stimulation for lower-limb prosthesis (Experimental)
  Interventions: Procedure: Peripheral Nerve Stimulation
- Spinal cord stimulation for upper-limb prosthesis (Experimental)
  Interventions: Procedure: Spinal cord stimulation
- Spinal cord stimulation for lower-limb prosthesis (Experimental)
  Interventions: Procedure: Spinal cord stimulation
- Dorsal root ganglion stimulation for upper-limb prosthesis (Experimental)
  Interventions: Procedure: Dorsal Root Ganglion Stimulation
- Experimental: Dorsal root ganglion stimulation for lower-limb prosthesis (Experimental)
  Interventions: Procedure: Dorsal Root Ganglion Stimulation
- Motor Cortex Stimulation for upper-limb prosthesis (Experimental)
  Interventions: Procedure: Motor Cortex Stimulation
- Motor Cortex Stimulation for lower-limb prosthesis (Experimental)
  Interventions: Procedure: Motor Cortex Stimulation

INTERVENTIONS:
Procedure: Peripheral Nerve Stimulation — Peripheral Nerve Stimulation (PNS) is a neuromodulation technique used to treat chronic pain. The procedure starts with a preoperative assessment, including imaging to identify the target peripheral nerve. Under local anesthesia, a thin, insulated electrode is implanted near the nerve, usually with the help of fluoroscopic or ultrasound guidance for precision.
  Arms: Peripheral nerve stimulation for lower-limb prosthesis; Peripheral nerve stimulation for upper-limb prosthesis
Procedure: Spinal cord stimulation — Spinal Cord Stimulation (SCS) is a neuromodulation that involves the implantation of a device that delivers electrical impulses to the spinal cord through an electrode placed in the epidural space. The stimulation alters pain signals before they reach the brain, effectively masking or reducing the sensation of pain.
  Arms: Spinal cord stimulation for lower-limb prosthesis; Spinal cord stimulation for upper-limb prosthesis
Procedure: Dorsal Root Ganglion Stimulation — Dorsal Root Ganglion Stimulation (DRGS) is a targeted neuromodulation technique for managing chronic pain. The procedure begins with a thorough preoperative assessment, including imaging to locate the specific dorsal root ganglion (DRG) associated with the pain. Under local anesthesia, a small electrode is implanted near the DRG. This is done through a minimally invasive procedure, often guided by fluoroscopy or CT imaging to ensure precise placement.
  Arms: Dorsal root ganglion stimulation for upper-limb prosthesis; Experimental: Dorsal root ganglion stimulation for lower-limb prosthesis
Procedure: Motor Cortex Stimulation — Motor Cortex Stimulation (MCS) is a neuromodulation technique that involves the surgical implantation of electrodes over the motor cortex, typically targeting the precentral gyrus, to deliver electrical stimulation. The procedure involves placing an electrode grid or strip on the dura mater overlying the motor cortex, which is identified via neuroimaging techniques such as functional MRI or neuronavigation. Once implanted, the electrodes are connected to an implanted pulse generator (IPG), which delivers adjustable electrical impulses.
  Arms: Motor Cortex Stimulation for lower-limb prosthesis; Motor Cortex Stimulation for upper-limb prosthesis

SUMMARY:
This clinical trial is designed to assess the effectiveness of advanced neuromodulation techniques in reducing phantom limb pain by improving sensory feedback in bionic prostheses. The study will explore the use of Peripheral Nerve Stimulation to evaluate their impact on pain relief and sensory restoration. The trial aims the development of neuroprostheses that can provide sensory feedback through stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Amputation of the upper limb at the level of the forearm or upper arm, or amputation of the lower limb at the level of the lower leg or thigh.
* Age between 18 and 65 years.
* Duration since amputation is at least 6 months.
* Presence of persistent chronic pain syndrome rated between 4 and 10 on the Visual Analog Scale (VAS).
* Absence of pregnancy at the time of implantation, confirmed by a pregnancy test (for female participants only).
* Signed consent to participate in the study.

Exclusion Criteria:

* Presence of severe somatic pathology that hinders surgical treatment and participation in the study.
* Presence of psychiatric disorders (including a history of), severe depression, suicidal tendencies, or a history of suicide attempts.
* Presence of severe orthopedic deformity in the limb above the level of amputation.
* History of cancer.
* History of epilepsy.
* Complicated traumatic brain injury (TBI) or a history of stroke.
* Inability to undergo electrostimulation due to other somatic pathology.
* Purulent-septic pathology.
* Drug addiction (including a history of).
* Congenital anomaly of upper limb development.
* Anomalies in the development of the central and peripheral nervous systems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
VAS | up to 4 months
  The Visual Analog Scale (VAS) is a 10 cm line used to measure pain intensity. One end of the line represents "no pain," while the other end signifies "worst possible pain." The line can be either horizontal or vertical.
SF-36 | up to months
  The questionnaire consists of 36 items grouped into eight scales: physical functioning, role limitations due to physical health, bodily pain, general health, vitality, social functioning, emotional well-being, and mental health. Each scale ranges from 0 to 100, where 100 represents full health. Higher scores indicate better quality of life, with two summary measures: physical and mental well-being.
DN 4 | Up to 6 months
  The DN4 (Douleur Neuropathique 4) questionnaire is a diagnostic tool designed to identify neuropathic pain, caused by nerve damage. It includes 10 items divided into two sections. The first part consists of seven questions that assess the patient's pain symptoms, such as burning, tingling, electric shocks, or numbness. The second part involves a clinical examination where the physician tests for reduced sensitivity to touch and pinprick, as well as pain response to light brushing. Each item is scored with 1 point for "Yes" and 0 for "No." A total score of 4 or higher indicates a high probability of neuropathic pain.

SECONDARY OUTCOMES:
Sensory threshold change | At least three measurements. 1 - First week after implantation, 2 - Up to three months after implantation, 3 - Up to five months after implantation
  In this task, the minimal amplitude of stimulation required to evoke a sensory response is experimentally determined. Numbers 1 and 2 appear on the screen, and at the moment one of the numbers appears, stimulation is simultaneously activated. The participant's task is to identify when the stimulation occurred and to input their response using the keyboard. After completing the task, a psychophysical curve will be computed, and the amplitude value that yields an accuracy of 0.75 will be used.
Agency | Up to 6 months
  Self-report questionnaires where participants rate their sense of agency over the prosthesis during tasks. It uses 0 to 10 scale, where 0 means lower agency and 10 means higher agency
Embodiment | Up to 6 months
  Throughout the study, participants will be asked to complete questionnaires assessing the degree of embodiment of the prosthesis. Since during the experimental sessions, feedback from the prosthesis is projected onto the phantom limb, the research team anticipates observing a transfer effect from the phantom limb to the robotic hand. The degree of this transfer will be evaluated using the Embodiment questionnaires for both upper and lower limbs.
  Embodiment uses scale from -9 to 9; -9 means "No embodiment" and 9 means "High embodiment".
Pain detect | Up to 6 months
  The questionnaire is intended for completion by a physician and combines a pain distribution diagram with a visual analog scale (VAS) and a section focused on identifying spontaneous and triggered neuropathic pain symptoms. It also assesses the nature of pain using the diagram, categorizing it as constant, episodic, or constant with episodes, among others. The questionnaire comprehensively reflects all possible pain parameters, allowing for clear tracking of pain dynamics over time.
  The total score ranges from -1 to 38. Based on this score:
  ≤ 12: Neuropathic pain is unlikely. 13-18: The result is ambiguous; further assessment may be needed.
  ≥ 19: Neuropathic pain is likely.
Hospital Anxiety and Depression Scale (HADS) | Up to 6 months
  The Hospital Anxiety and Depression Scale (HADS) is a widely used screening tool designed to assess anxiety and depression levels in patients in non-psychiatric hospital settings. It consists of 14 items, divided into two subscales: seven questions assess anxiety (HADS-A) and seven assess depression (HADS-D). The items focus on emotional and cognitive symptoms rather than physical symptoms, making it suitable for patients with medical conditions. Each item is scored on a scale of 0 to 3, with total scores for each subscale ranging from 0 to 21. A score of 8 or more on either subscale suggests the presence of anxiety or depression. The HADS is valued for its simplicity and reliability in clinical and research settings.
Ownership | Up to 6 months
  Self-report questionnaires where participants rate their sense of ownership over the prosthesis during tasks. It uses 0 to 10 scale, where 0 means lower agency and 10 means higher agency

OTHER OUTCOMES:
Object detection | Up to 6 months
  In a task that requires distinguishing object sizes using feedback from a prosthetic hand grasps objects made of different materials, of varying shapes, or of the same shape but with different diameters.
Visual-motor integration | Up to 4 months
  The participant's task is to transport an object within designated zones using their prosthesis. In each trial, the target zone is randomly determined, and the participant must move the object to this zone as quickly and accurately as possible. The experimental conditions include sessions where neuroprosthetic feedback is active and others where the system is disabled. During the task, the participant wears eye tracking glasses. Investigators measure the number and duration of fixations on the prosthesis.
Value of sensory discrimination | Up to once in two weeks
  Value of sensory discrimination is measured as Accuracy of Object Recognition. In this task, patients distinguish object sizes using feedback from stimulation through a prosthetic hand. The hand grasps objects made from various materials, with different shapes, or the same shape but different diameters. Concurrently, signals from the prosthetic sensors are translated into patterns of electrical stimulation. When the patient initiates a grasp, changes in the sensor signals result in adjustments to the amplitude of the neurostimulation. The patient's goal is to identify the properties of the objects based solely on the neurostimulation signals, while visual and auditory cues are blocked with a mask and headphones. It is expected that as patients adapt to the prosthetic system, their performance in recognizing objects will improve over time.
Grasping surface differentiation | Up to 6 months
  In this task, the participant is presented with three identical objects, each assigned to one of three classes: (1) a non-tactile object, (2) a tactile object, and (3) a highly tactile object. At the start of each trial, the object classes are randomly reassigned. The distinction between the classes is that, upon touching an object of class (1) with the prosthesis, the participant receives no feedback; touching a class (2) object triggers low-amplitude stimulation, and a class (3) object triggers high-amplitude stimulation. During the trial, the participant uses the prosthesis to examine each object and determine which one belongs to class 2. As a final measurement investigators take the accuracy in this task.
Sensory discrimination ability | up to 4 months
  In a task requiring the discrimination of objects using feedback from stimulation, the prosthetic hand grasps objects made of different materials, varying shapes, or identical shapes but different diameters. Simultaneously, signals from the prosthetic sensors are transformed into patterns of electrical stimulation. When the patient initiates a grasp, changes in the sensor data result in alterations in the amplitude of neurostimulation. The patient's task is to determine the properties of the objects based on the signals from neurostimulation, while other sources of information-visual and auditory-are blocked using a bandage and headphones. It is expected that over time, as patients adapt to the prosthetic system, their performance in this task will improve. The final measure is an accuracy of discrimination computed as correct responses divided bu number of trials
Clothespin relocation task | Up to 6 months
  The test requires at least two movements in the prosthesis: hand opening-closing and wrist supination-pronation. In the test, the subject stands with the prosthetic arm lowered and elbow extended. They must move three red clips from a horizontal to a vertical rod and back, using a Rolyan Graded Pinch Exerciser. The feet must remain on the floor, and the time to complete the task is recorded.
Fragile objects | Up to 6 months
  In this task, the participant is asked to move a fragile object from one area to another using a neuroprosthetic system. The challenge lies in the fact that moving the fragile object requires precise motor control, as excessive pressure may break it. The participant must move the object as many times as possible within a 1-minute window.
Sensory feedback in a virtual prosthesis | Up to 6 months
  In this paradigm, the participant controls a prosthesis in VR. Myographic sensors control various grasps of the virtual prosthesis, and when the prosthetic avatar touches virtual objects, a neurostimulation-based feedback system is activated. The quality of prosthesis control is estimated
Treadmill | Up to 6 months
  In this task, the participant takes a fixed-duration walk on a treadmill at a set speed while connected to a motion capture system and spirometry. The walk includes two modes: with and without feedback. The leg prosthesis feedback system operates via signals from a smart insole, modulating stimulation based on signal changes. Gait patterns from sessions with and without feedback will be compared, and changes in respiratory patterns are also expected between the two modes.
Standing Surface Discrimination | Up to 6 months
  In this task, a smart insole equipped with a pressure sensor system is connected to the leg prosthesis. Using transformation of the sensor data, the neurostimulation signal is modulated to encode different patterns of pressure applied to the insole. The patient's objective is to learn to distinguish between various surfaces in contact with the insole. This test assesses the sensory discrimination capabilities of the sensory-enabled lower limb prosthesis.
Staircase test | Up to 6 months
  The test aims to compare functional mobility when ascending and descending stairs with and without feedback. The time taken to climb one flight of stairs, turn on the landing, and descend is measured. Multiple attempts are given with a 2-minute rest between them, and the best result is recorded.
OPUS (Orthotics and Prosthetics User Survey) | Up to 6 months
  OPUS (Optimal Patient Utilization System) is a clinical decision support tool designed to enhance patient care through improved resource management and treatment efficiency. It utilizes advanced algorithms and data analytics to optimize patient scheduling, treatment pathways, and staff allocation within healthcare facilities. By analyzing patient demographics, medical history, and treatment outcomes, OPUS helps clinicians make informed decisions about resource allocation and care delivery. The system aims to reduce wait times, streamline operations, and improve overall patient satisfaction. Additionally, OPUS provides real-time feedback and reporting capabilities, enabling healthcare providers to monitor performance metrics and identify areas for improvement, ultimately enhancing the quality of care.
PEQ (Prosthesis Evaluation Questionnaire) | Up to 6 months
  The Prosthesis Evaluation Questionnaire (PEQ) is a standardized assessment tool designed to evaluate the functional and psychosocial outcomes of individuals using prosthetic devices. Comprising various domains, the PEQ addresses aspects such as mobility, activity level, and quality of life, allowing users to report their experiences and satisfaction with their prosthesis. The questionnaire includes specific items that gauge the user's perception of their prosthetic limb's comfort, functionality, and impact on daily activities. PEQ ranges from 0 to 100: 0 indicates the worst possible outcome (e.g., "not at all satisfied") and 100 indicates the best possible outcome (e.g., "completely satisfied").
Box and blocks | Up to 6 months
  The setup includes an open box with a divider, 150 wooden blocks, and a timer. The participant, seated at a table, has 60 seconds to move as many blocks as possible, one at a time, over the divider using one hand.
TMS induced muscle potentials | Up to 6 months
  To assess the functional state of motor nerves in the amputated limb, transcranial magnetic stimulation (TMS) will be used. A TMS stimulator, consisting of one or two electromagnetic coils, will be placed over the motor cortex, while an electromyographic (EMG) electrode will be positioned over the target muscle of the amputated limb. A current pulse through the TMS coils will induce currents in the motor cortex, activating it and eliciting motor-evoked potentials (MEPs) in the target muscle. Delays and EMG potential profiles will inform on motor nerve function and the suitability of neuromodulation, as well as the therapeutic effects of TMS for phantom limb pain relief.

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Federal Center of Brain Research and Neurotechnologies of the Federal Medical Biological Agency of Russia, Moscow
  - Far Eastern Federal University, Moscow